CLINICAL TRIAL: NCT01271725
Title: LUX-Breast 2; An Open Label, Phase II Trial of Afatinib (BIBW 2992) in Patients With Metastatic HER2-overexpressing Breast Cancer Failing HER2-targeted Treatment in the Neoadjuvant and/or Adjuvant Treatment Setting
Brief Title: LUX-Breast 2; Afatinib in HER2 (Human Epidermal Growth Factor Receptor)-Treatment Failures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.98; 2010-021945-29 (EudraCT Number)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Afatinib; Paclitaxel

ARMS (3):
- Afatinib 40mg once daily (OD) (Experimental): Patient to receive afatinib monotherapy at a dose of 40 mg/d until progression of their disease
  Interventions: Drug: Afatinib 40mg once daily (OD)
- Paclitaxel 80 mg/m2 weekly (Experimental): Patients to additionally receive paclitaxel at a dose of 80 mg/m2 weekly on disease progression on afatinib monotherapy
  Interventions: Drug: Paclitaxel 80 mg/m2 weekly
- Vinorelbine 25 mg/m2 weekly (Experimental): Patients to additionally receive vinorelbine at a dose of 25 mg/m2 weekly on disease progression on afatinib monotherapy
  Interventions: Drug: Vinorelbine 25 mg/m2 weekly

INTERVENTIONS:
Drug: Vinorelbine 25 mg/m2 weekly — Patients to additionally receive vinorelbine at a dose of 25 mg/m2 weekly on disease progression on afatinib monotherapy
  Arms: Vinorelbine 25 mg/m2 weekly
Drug: Afatinib 40mg once daily (OD) — Patient to receive afatinib monotherapy at a dose of 40 mg/d until progression of their disease
  Arms: Afatinib 40mg once daily (OD)
Drug: Paclitaxel 80 mg/m2 weekly — Patients to additionally receive paclitaxel at a dose of 80 mg/m2 weekly on disease progression on afatinib monotherapy
  Arms: Paclitaxel 80 mg/m2 weekly

SUMMARY:
The general aim of this study is to investigate the efficacy and safety of afatinib (BIBW 2992) alone and in combination with weekly paclitaxel or weekly vinorelbine (in patients who progress on afatinib monotherapy within this trial) as treatment in patients with HER2-overexpressing, metastatic breast cancer, who failed HER2-targeted treatment in the neoadjuvant or adjuvant setting

ELIGIBILITY:
Inclusion criteria:

1. Female patients >=18 years with proven diagnosis of HER2-overexpressing, histologically confirmed breast cancer
2. Stage IV metastatic disease
3. At least one measurable lesion according to RECIST 1.1 (Response Evaluation Criteria for Solid Tumours version 1.1). Skin, bone and brain lesions are considered non-target lesions
4. Must have failed or progressed on either trastuzumab or lapatinib or trastuzumab and lapatinib treatment in the neoadjuvant and/or adjuvant setting

Exclusion criteria:

1. Prior first line therapy for metastatic breast cancer
2. Known pre-existing interstitial lung disease
3. Active brain metastases
4. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to trial treatment.
5. Cardiac left ventricular function with resting ejection fraction of less than 50%.
6. Prior treatment with Epidermal Growth Factor Receptor (EGFR)/HER2-targeted small molecules or antibodies other than trastuzumab and lapatinib in the neoadjuvant or adjuvant setting
7. Prior treatment with paclitaxel in the past 12 months
8. Must not have received prior vinorelbine treatment - Further exclusion criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-05-24 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (27):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- India (6):
  - Sujan Surgical Cancer Hospital, Amravati
  - Tata Memorial Hospital, Maharashtra
  - Curie Manavata Cancer Centre, Maharashtra
  - Central India Cancer Research Institute, Nagpur
  - Ruby Hall Clinic, Pune
  - Regional Cancer Center, Thiruvananthapuram
- University Clinical Center, Gdansk, Gdansk, Poland
- Russia (8):
  - St.Auton.Heal.Inst."Rep.Clin.Onc.Disp.of MoH of Rep. Tatarstan", Kazan'
  - Clinical Oncology Dispensary No. 1, Dept. Chemotherapy, Krasnodar
  - N.A. Semashko Central Clinical Hospital, Moscow, Moscow
  - SBIH of Stavropol territory "Pyatigorsk Oncol. Dispensary", Pyatigorsk
  - SBIH "Samara Regional Clinical Oncol. Dispensary", Samara, Samara
  - GUZ "Oncological Dispesary #2", Sochi
  - Stavropol Regional Clin. Oncology Dispensary Dept. Oncology, Stavropol
  - Yaroslavl Regional Clinical Oncology Hosp. Dept.Chemotherapy, Yaroslavl
- Taiwan (6):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Koo Foundation Sun Yet-Sen Cancer Center, Taipei
  - Taipe Veterans General Hospital, Taipei
- United Kingdom (4):
  - North Devon District Hospital, Barnstaple
  - Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Royal Devon and Exeter Hospital, Exeter
  - Charing Cross Hospital, London

REFERENCES:
- [Derived] Hickish T, Mehta A, Liu MC, Huang CS, Arora RS, Chang YC, Yang Y, Vladimirov V, Jain M, Tsang J, Pemberton K, Sadrolhefazi B, Jin X, Tseng LM. Afatinib alone and in combination with vinorelbine or paclitaxel, in patients with HER2-positive breast cancer who failed or progressed on prior trastuzumab and/or lapatinib (LUX-Breast 2): an open-label, multicenter, phase II trial. Breast Cancer Res Treat. 2022 Apr;192(3):593-602. doi: 10.1007/s10549-021-06449-4. Epub 2022 Feb 9. PMID 35138529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, multinational, phase-II trial of Afatinib (BIBW 2992) in patients with metastatic human epidermal growth factor receptor (HER2) - overexpressing breast cancer failing HER2 - targeted treatment in the neoadjuvant and/or adjuvant treatment setting
Pre-assignment Details: All subjects were screened for eligibility. It was not planned to compare efficacy of the combination therapies "Afatinib and Paclitaxel or Afatinib and Vinorelbine" as the study was stopped prematurely and the patient number in both treatment groups is not significant. However, for safety reporting both combination therapy are reported separately
Groups:
- Afatinib Monotherapy: Patient received Afatinib monotherapy orally once daily at a dose of 40 milligram (mg) film-coated tablets until progression of their disease, unacceptable adverse events or other reason necessitating withdrawal. Patients could have dose reduced if 40 mg was not tolerated.
- Afatinib and Paclitaxel or Vinorelbine Combination Therapy: Patient received Afatinib monotherapy orally once daily at a dose of 40 mg film-coated tablets until progression of their disease, unacceptable adverse events or other reason necessitating withdrawal (Patients could have dose reduced if 40 mg was not tolerated) and 80 mg/square meter (m2) Paclitaxel concentrate for intravenous infusion or 25 mg/m2 Vinorelbine concentrate for intravenous infusion once weekly starting after treatment failure on afatinib monotherapy
Period: Part A
Arm/Group | Afatinib Monotherapy | Afatinib and Paclitaxel or Vinorelbine Combination Therapy
Started | 74 (Started are the treated patients) | 0
Completed | 39 | 0
Not Completed | 35 | 0
Not completed — Progressive disease according to RECIST | 8 | 0
Not completed — Clinical signs/symptoms of progression | 2 | 0
Not completed — Other Adverse Event | 8 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 12 | 0
Not completed — Other than specified | 3 | 0
Not completed — Protocol Violation | 1 | 0
Period: Part B
Arm/Group | Afatinib Monotherapy | Afatinib and Paclitaxel or Vinorelbine Combination Therapy
Started | 0 | 39
Completed | 0 | 27 (Patient deemed to have completed the trial once they showed progressive disease according to RECIST)
Not Completed | 0 | 12
Not completed — Other than specified | 0 | 2
Not completed — Clinical signs/symptoms of progression | 0 | 2
Not completed — Other Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 6

BASELINE CHARACTERISTICS:
Population: The treated set for monotherapy comprised all patients who received at least 1 dose of afatinib. The treated set for combination therapy comprised all patients who received at least 1 dose of each of afatinib and paclitaxel, or of afatinib and vinorelbine.
Arm/Group | Afatinib Monotherapy
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented.
  Years | 51.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female.
  Participants
    Female | 74
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not captured in this trial
  Participants
    American Indian or Alaska Native | 0
    Asian | 47
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 27
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR) Assessed by Response Evaluation Criteria in Solid Tumours Version (RECIST) 1.1
Description: Objective response according to RECIST v1.1. Best overall response of confirmed complete response (CR) or confirmed partial response (PR) recorded since first administration of trial medication and until the earliest of disease progression, death or start of next treatment in each part separately. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by Magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR. Percentage of participants with OR along with exact 95% Confidence Interval by Clopper and Pearson is presented.
Time Frame: From the initial dose of study drug until 28 days after end of the treatment period, up to 1562 days
Population: The treated set for monotherapy comprised all patients who received at least 1 dose of afatinib. Treated set for combination therapy comprised all patients who received at least 1 dose of each of afatinib and paclitaxel or of afatinib and vinorelbine. It was not planned to compare between the two types of combination therapies hence arm is combined
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib Monotherapy | Afatinib and Paclitaxel or Vinorelbine Combination Therapy
Number analyzed (Participants) | 74 | 39
Percentage of participants | 18 [10 to 28] | 31 [17 to 48]

2. Secondary Outcome: Best Overall Response According to RECIST v1.1 (With Confirmation)
Description: Best overall response was assessed according to RECIST version 1.1 and was calculated relative to the baseline of each respective part .Percentage of participants with best overall response along with exact 95% Confidence Interval by Clopper and Pearson is presented. Best overall response was defined as the best response recorded at any time from the first administration of drug to the End of Treatment (EOT). As Per RECIST v1.1 for target lesions and assessed by Magnetic resonance imaging (MRI): Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least 30% decrease in the sum of the longest diameter of target lesions; progression, at least 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: From the initial dose of study drug until 28 days after end of the treatment period, up to 1562 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib Monotherapy | Afatinib and Paclitaxel or Vinorelbine Combination Therapy
Number analyzed (Participants) | 74 | 39
Percentage of participants
  Complete response (CR) | 1 [0 to 7] | 0 [0 to 9]
  Partial response (PR) | 16 [9 to 27] | 31 [17 to 48]
  Stable disease (SD) | 45 [33 to 57] | 46 [30 to 63]
  Progressive disease | 28 [19 to 40] | 10 [3 to 24]
  Not evaluable | 9 [4 to 19] | 13 [4 to 27]

3. Secondary Outcome: Best Overall Response According to RECIST v1.1 (Regardless of Confirmation)
Description: Best overall response was assessed according to RECIST version 1.1 and was calculated relative to the baseline of each respective part (without clinical disease assessment) .Percentage of participants with best overall response along with exact 95% Confidence Interval by Clopper and Pearson is presented. Best overall response was defined as the best response recorded at any time from the first administration of drug to the End of Treatment (EOT). As Per RECIST v1.1 for target lesions and assessed by Magnetic resonance imaging (MRI): Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least 30% decrease in the sum of the longest diameter of target lesions; progression, at least 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: From the initial dose of study drug until 28 days after end of the treatment period, up to 1562 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib Monotherapy | Afatinib and Paclitaxel or Vinorelbine Combination Therapy
Number analyzed (Participants) | 74 | 39
Percentage of participants
  Complete response (CR) | 1 [0 to 7] | 0 [0 to 9]
  Partial response (PR) | 19 [11 to 30] | 44 [28 to 60]
  Stable disease (SD) | 42 [31 to 54] | 33 [19 to 50]
  Progressive disease | 28 [19 to 40] | 10 [3 to 24]
  Not evaluable | 9 [4 to 19] | 13 [4 to 27]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the time from the drug start date to the date of 1st disease progression or death for monotherapy and 2nd disease progression or death from the drug start date of the combination therapy for combination therapy'. Median is calculated from the Kaplan-Meier curve.
Time Frame: From drug start date in monotherapy to 1st disease progression and drug start date in combination therapy to 2nd disease progression
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Afatinib Monotherapy | Afatinib and Paclitaxel or Vinorelbine Combination Therapy
Number analyzed (Participants) | 74 | 39
Days | 86.0 [72.0 to 127.0] | 135.0 [95.0 to 224.0]

5. Secondary Outcome: Duration of Objective Response According to RECIST v1.1
Description: Duration of objective response, defined as the time from first objective response to the time of progression or death. (regardless of confirmation). As Per RECIST v1.1 for target lesions and assessed by Magnetic resonance imaging (MRI): Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least 30% decrease in the sum of the longest diameter of target lesions; progression, at least 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: From the first objective response to the time of progression or death, up to 1562 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Afatinib Monotherapy | Afatinib and Paclitaxel or Vinorelbine Combination Therapy
Number analyzed (Participants) | 74 | 39
Days | 168.5 [85.0 to 253.0] | 125.0 [73.0 to 505.0]

6. Secondary Outcome: Percentage of Patients With Highest Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 Grade of 3 or Higher
Description: Percentage of patients with highest common terminology criteria for adverse events (CTCAE) version 3.0 Grade of 3 or higher.
Time Frame: From the initial dose of study drug until 28 days after end of the treatment period, up to 1562 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Groups:
- Afatinib and Vinorelbine Combination Therapy: Patient received Afatinib monotherapy orally once daily at a dose of 40 mg film-coated tablets until progression of their disease, unacceptable adverse events or other reason necessitating withdrawal (Patients could have dose reduced if 40 mg was not tolerated) and 25 mg/m2 Vinorelbine concentrate for intravenous infusion once weekly starting after treatment failure on afatinib monotherapy
- Afatinib and Paclitaxel Combination Therapy: Patient received Afatinib monotherapy orally once daily at a dose of 40 mg film-coated tablets until progression of their disease, unacceptable adverse events or other reason necessitating withdrawal (Patients could have dose reduced if 40 mg was not tolerated) and 80 mg/square meter (m2) Paclitaxel concentrate for intravenous infusion once weekly starting after treatment failure on afatinib monotherapy
Arm/Group | Afatinib Monotherapy | Afatinib and Vinorelbine Combination Therapy | Afatinib and Paclitaxel Combination Therapy
Number analyzed (Participants) | 74 | 13 | 26
Percentage of participants | 43 | 62 | 65

7. Secondary Outcome: Change From Baseline to End of Treatment in Systolic Blood Pressure (SBP)
Description: Change from baseline to end of treatment in systolic blood pressure (SBP).
Time Frame: Baseline and End of treatment period, up to 1562 days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Afatinib Monotherapy | Afatinib and Vinorelbine Combination Therapy | Afatinib and Paclitaxel Combination Therapy
Number analyzed (Participants) | 74 | 13 | 26
Millimeter of mercury (mmHg) | -1.2 (17.9) | -1.0 (15.1) | -3.7 (12.1)

8. Secondary Outcome: Change From Baseline to End of Treatment in Diastolic Blood Pressure (DBP)
Description: Change from baseline to end of treatment in diastolic blood pressure (DBP).
Time Frame: Baseline and End of treatment period, up to 1562 days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Afatinib Monotherapy | Afatinib and Vinorelbine Combination Therapy | Afatinib and Paclitaxel Combination Therapy
Number analyzed (Participants) | 74 | 13 | 26
Millimeter of mercury (mmHg) | -1.8 (12.0) | 1.9 (10.7) | -1.6 (10.0)

9. Secondary Outcome: Number of Patient With Possibly Clinically Significant (PCS) Laboratory Values
Description: Number of patient with possibly clinically significant (PCS) laboratory values by functional group (haematology, differentials, coagulation, electrolytes, enzymes, and substrates). Acronyms Used: Prothrombin time-International normalized ratio (PT-INR), Alanine aminotransferase/Glutamic pyruvic transaminase (ALT/GPT) Serum glutamic pyruvic transaminase (SGPT), Aspartate aminotransferase/Glutamic-oxaloacetic transaminase (AST/GOT) Serum glutamic-oxaloacetic transaminase (SGOT)
Time Frame: From the initial dose of study drug until 28 days after end of the treatment period, up to 1562 days
Population: The treated set for monotherapy comprised all patients who received at least 1 dose of afatinib. Number Analyzed are the patients with no possible clinically significant abnormality at baseline. Treated set for combination therapy comprised all patients who received at least 1 dose of each of afatinib and paclitaxel, or of afatinib and vinorelbine.
Measure: Number; unit: Participants
Arm/Group | Afatinib Monotherapy | Afatinib and Vinorelbine Combination Therapy | Afatinib and Paclitaxel Combination Therapy
Number analyzed (Participants) | 74 | 13 | 26
Participants
  Haematology - Haemoglobin (low): number analyzed (Participants) | 71 | 13 | 26
  Haematology - Haemoglobin (low) | 9 | 5 | 17
  Haematology - White blood cell count (low): number analyzed (Participants) | 71 | 13 | 26
  Haematology - White blood cell count (low) | 5 | 9 | 13
  Haematology - Platelets (low): number analyzed (Participants) | 71 | 13 | 26
  Haematology - Platelets (low) | 2 | 0 | 1
  Differentials, automatic - Neutrophils (low): number analyzed (Participants) | 71 | 13 | 26
  Differentials, automatic - Neutrophils (low) | 1 | 10 | 12
  Coagulation - PT-INR (high): number analyzed (Participants) | 63 | 13 | 25
  Coagulation - PT-INR (high) | 1 | 0 | 0
  Electrolytes - Potassium (low): number analyzed (Participants) | 70 | 13 | 26
  Electrolytes - Potassium (low) | 3 | 0 | 3
  Electrolytes - Potassium (high): number analyzed (Participants) | 70 | 13 | 26
  Electrolytes - Potassium (high) | 2 | 0 | 0
  Electrolytes - Magnesium (low): number analyzed (Participants) | 63 | 12 | 25
  Electrolytes - Magnesium (low) | 0 | 0 | 1
  Enzymes - AST/GOT SGOT (high): number analyzed (Participants) | 70 | 13 | 26
  Enzymes - AST/GOT SGOT (high) | 8 | 0 | 2
  Enzymes - ALT/GPT SGPT (high): number analyzed (Participants) | 71 | 13 | 26
  Enzymes - ALT/GPT SGPT (high) | 6 | 3 | 4
  Enzymes - Alkaline phosphatase (high): number analyzed (Participants) | 71 | 13 | 26
  Enzymes - Alkaline phosphatase (high) | 6 | 1 | 2
  Substrates - Creatinine (high): number analyzed (Participants) | 71 | 13 | 26
  Substrates - Creatinine (high) | 0 | 0 | 1
  Substrates - Bilirubin, total (high): number analyzed (Participants) | 71 | 13 | 26
  Substrates - Bilirubin, total (high) | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: From the initial dose of study drug until 28 days after end of the treatment period, up to 1562 days
Description: Safety analyses were performed for monotherapy and combination therapy separately using the respective treated sets.The treated set for monotherapy comprised all patients who received at least 1 dose of afatinib. The treated set for combination therapy comprised all patients who received at least 1 dose of each of afatinib and paclitaxel, or of afatinib and vinorelbine.
Arm/Group | Afatinib Monotherapy | Afatinib and Vinorelbine Combination Therapy | Afatinib and Paclitaxel Combination Therapy
All-Cause Mortality (participants affected / at risk) | 6/74 | 1/13 | 5/26
Serious Adverse Events (participants affected / at risk) | 18/74 | 5/13 | 10/26
Other Adverse Events (participants affected / at risk) | 67/74 | 13/13 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Monotherapy (N=74) | Afatinib and Vinorelbine Combination Therapy (N=13) | Afatinib and Paclitaxel Combination Therapy (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Asthenia (General disorders) | 3 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 2
Brain oedema (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Device leakage (Product Issues) | 1 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Monotherapy (N=74) | Afatinib and Vinorelbine Combination Therapy (N=13) | Afatinib and Paclitaxel Combination Therapy (N=26)
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 13
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 1 | 9 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 3 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 3
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 50 | 3 | 9
Haemorrhoids (Gastrointestinal disorders) | 3 | 1 | 2
Mouth ulceration (Gastrointestinal disorders) | 8 | 2 | 2
Nausea (Gastrointestinal disorders) | 9 | 1 | 4
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2 | 4
Asthenia (General disorders) | 5 | 2 | 7
Fatigue (General disorders) | 7 | 0 | 5
Mucosal inflammation (General disorders) | 15 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 2
Pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 4 | 1 | 2
Ulcer (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 4 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2
Paronychia (Infections and infestations) | 9 | 2 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 3
Viral infection (Infections and infestations) | 0 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0 | 4
Aspartate aminotransferase (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 4 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 2
Blood uric acid increased (Investigations) | 2 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 2 | 1
Weight decreased (Investigations) | 10 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 1
Headache (Nervous system disorders) | 7 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 4
Insomnia (Psychiatric disorders) | 1 | 0 | 3
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 4 | 1 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 37 | 3 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Phlebitis (Vascular disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Enrollment of patients into the afatinib and vinorelbine combination option was stopped prematurely following a benefit-risk analysis in other trial. Any patients who were already benefiting from this combination were allowed to continue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-10-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT01271725/SAP_000.pdf
  • Study Protocol (2013-06-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT01271725/Prot_001.pdf